CLINICAL TRIAL: NCT05483790
Title: Enhancing Latent Cognitive Capacity in Community-Dwelling Older Adults With or At-Risk for Mild Cognitive Impairment（MCI): a RCT Study
Brief Title: The Effects of Multidomain Non-pharmacological Interventions on the Elderly With or Without Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Collaborators: School of Public Health，Fudan University (Unknown); Medicine-Mental Health Center of Minhang District (Unknown); Xinzhuang Community Health Service Center (Unknown)
Responsible Party: Principal Investigator, Huang Yanyan, Professor (Department of General Medicine, Department of Geriatrics), Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017YFC1310504
Record Dates: First submitted 2022-07-24; First posted 2022-08-02 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Mild Cognitive Impairment; The Cognitive Normal Elderly
Keywords: mild cognitive impairment; the elderly; non-pharmacological intervention; cognitive function; magnetic resonance imaging; randomized controlled trial
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: the intervention group and the control group
Who Masked: Outcomes Assessor
Masking Description: single-blinding was pursued as much as possible: group allocation was not actively disclosed to participants, they were advised not to discuss the intervention during testing sessions, opportunities for between-group interactions were restricted, and outcome assessors were blinded to allocation and were not involved in the intervention activities.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multidomain intervention (Experimental): The interventions were conducted for 6-week training phase and 6-week maintenance phase. Including cognitive training, physical exercise, healthy lifestyle education, and computerized interaction training. The multimodal intervention program included the in-person training course (90-minute, once per week for 6 weeks), computerized interaction training (30-minute, 3 times per week for 6 weeks), and homework (30-minute, every day for 12 weeks).
  Interventions: Behavioral: the multimodal intervention
- the control (No Intervention): Throughout the 6-week training phase and 6-week maintenance period, the control group only received 30-minute health education through booklets, home visits, or phone calls once every week.

INTERVENTIONS:
Behavioral: the multimodal intervention — The in-person training course included 25 minutescognitive training activities were conducted for , followed by a 15-minute healthy lifestyle education. After a 10-minute break, physical exercise training was administered for 15 minutes. Finally, 15 minutes wrap-up session.
  The cognitive training encompassed memory-related training and attention-related training. The physical exercise included finger exercises, elastic band exercises, Tai Chi/ Baduanjin with guidance. The healthy lifestyle education included guidance on nutrition, sleep, stress management, and mood adjustment by teaching problem-solving skills. Additionally, the intervention provided information and support to facilitate lifestyle changes and included discussions and practical exercises, such as tools for assessing dietary behavior.
  Arms: multidomain intervention

SUMMARY:
The study aiming to investigate the efficacy, safety, and potential mechanism of a multimodal intervention on cognitive function in individuals with MCI or the cognitive normal elderly living in a community. The recruited elderly aged 50-75 years with normal cognitive function or MCI will be divided into the intervention group or the control group randomly. The intervention group will be accepted a multidimensional non-pharmacological intervention (cognitive training, physical exercise, healthy lifestyle intervention, and computerized interaction training) while the control group receives health education. Sociodemographics will be collected before the intervention. comprehensive neuropsychological tests and MRI will be collected before and 6 weeks, 12 weeks, 3 months, 6 months, 12 months after the randomization respectively.

DETAILED DESCRIPTION:
This study is a 6-week training phase and 6-week maintenance phase randomized controlled trial, conducted at Xinzhuang Town, Minhang District, Shanghai, China.

All participants (control and intervention group) complete the data collection. Demographic data will be collected before intervention including age, sex, education, marriage, etc. A comprehensive cognitive assessment and MRI will be done before and 6 weeks, 12 weeks,3 months, 6 months, 12 months after the randomization respectively.

The intervention group receive four intervention components including cognitive training, physical exercise, healthy lifestyle intervention, and computerized cognitive training. a multimodal intervention program (with schedule) was conducted in the intervention group for 6-week training phase and 6-week maintenance, including cognitive training, physical exercise, healthy lifestyle education, and computerized interaction training. Throughout the 12-week period, the control group only received 30-minute health education through booklets, home visits, or phone calls once every week. The multimodal intervention program included the in-person training course (90-minute, once per week for 6 weeks), computerized interaction training (30-minute, 3 times per week for 6 weeks), and homework (30-minute, every day for 12 weeks).

The in-person training course started with a 10-minute period of reminiscence and discussion. Subsequently, cognitive training activities were conducted for 25 minutes, followed by a 15-minute healthy lifestyle education. After a 10-minute break, physical exercise training was administered for 15 minutes. Finally, participants summarized the all-training activities, either through writing or discussion, and planed their homework during a 15-minute wrap-up session.

The cognitive training encompassed memory-related training (i.e. picture recall, categorization, cueing, repetition, association, sentence formation, story construction, utilization of the Roman room method, face-name association, and verbalization to aid retention) and attention-related training (i.e. character-picture association, idiom-picture association, and spot-the-difference tasks were incorporated). The physical exercise included finger exercises, elastic band exercises, Tai Chi/ Baduanjin with guidance. The healthy lifestyle education included guidance on nutrition, sleep, stress management, and mood adjustment by teaching problem-solving skills, such as managing stressful life events and handling anger and frustration. Additionally, the intervention provided information and support to facilitate lifestyle changes and included discussions and practical exercises, such as tools for assessing dietary behavior.

The instructor-supervised, computer program-based computerized interaction training three times weekly included spatial cognition (i.e. participants manipulated identical cubes or two-dimensional figures in different orientations using a control handle), left and right brain balance tasks (i.e. replicating graphics from one computer screen to another using action tracking or screen touching technology), clock imitation exercises (i.e. participants mimicked the movements of hour and minute hands to match the time displayed on the computer screen), and automatic teller machine simulation (i.e. wherein participants performed transactions like cash withdrawals, money transfers, and balance checks using a computer interface similar to an ATM, while also recalling passwords and transaction amounts.

The every-day homework encompassed activities such as calligraphy practice (2 days per week) and physical exercise (the other 5 days per week). Participants were asked to complete their homework within approximately 30 minutes and share pictures or videos of their homework in a WeChat group each day, allowing for assessment of their adherence.

The trial is conducted by local health workers, who were trained by a team comprising neurologists and geriatrics experts from Huashan Hospital. The training manuals, demo videos, education resources (such as PowerPoint files and materials) and standardized health education study materials were also distributed to them.

The control group receives regular health advice weekly through brochures, home visits, or telephone calls during 6-week training phase and 6-week maintenance period, detail including (1) patients with cognitive impairment education: prevention from self-injury, falling injury, accidental injury, medication, lost and bad habits; (2) inmates or caregivers education; (3) cognitive impairment knowledge education; (4) prevention of cognitive dysfunction education. The intervention committee ensures that health education activities are consistent across sites and unlikely to increase physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥50 and ≤75 years, Male or Female
2. The resident elderly or those who have lived in the sampled community for more than 6 months
3. Be able to communicate with investigators and understand the questionnaire questions
4. More than 6 years of education
5. Mild cognitive impairment according to the Peterson criteria
6. Volunteer to participate in the study

Exclusion Criteria:

1. Individuals with neurological diseases
2. Cognitive decline due to other disorders (cerebrovascular disease, central nervous system infections, etc.)
3. Mental Disorders included in The Diagnostic and Statistical Manual of Mental Disorders of The American Psychiatric Association
4. Blindness, aphasia, or severe hearing impairment
5. History of myocardial infarction within the previous year, Unstable cardiac, renal, lung, liver or other severe chronic diseases
6. Coincident participation in another intervention trial
7. Using pharmacologic therapeutics for cognitive impairment.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
cognitive function assessed by the Mini-Mental State Examination (MMSE) | Before the intervention
  MMSE using the Chinese version revised by Zhang Mingyuan, the scale includes 30 items, including orientation, instantaneous memory, attention, computation, recall, language and visuospatial. The MMSE score ranges from 0 to 30 (30=best).
cognitive function assessed by the Mini-Mental State Examination (MMSE) | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  MMSE using the Chinese version revised by Zhang Mingyuan, the scale includes 30 items, including orientation, instantaneous memory, attention, computation, recall, language and visuospatial. The MMSE score ranges from 0 to 30 (30=best).

SECONDARY OUTCOMES:
memory function assessed by AVLT | Before the intervention
  Auditory Verbal Learning Test（AVLT）to rate immediate (sum of words recalled on the 5 learning trials) and delayed episodic verbal memory.
memory function assessed by AVLT | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  Auditory Verbal Learning Test（AVLT）to rate immediate (sum of words recalled on the 5 learning trials) and delayed episodic verbal memory.
memory function assessed by LMT | Before the intervention
  Logic memory test (LMT): which assesses memory for brief passages, similar to newspaper stories. Subjects were assessed on immediate recall and 30 minute interval for delayed recall, according to standard practice. Subjects were not instructed in advance that they would be re-tested on the story after a delay of 30 minutes.
memory function assessed by LMT | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  Logic memory test (LMT): which assesses memory for brief passages, similar to newspaper stories. Subjects were assessed on immediate recall and 30 minute interval for delayed recall, according to standard practice. Subjects were not instructed in advance that they would be re-tested on the story after a delay of 30 minutes.
executive function assessed by TMT-A | Before the intervention
  The trail marking test A (TMT-A): The TMT-A consisted of a standardized page on which the numbers 1 to 25 are scattered within circles, and the participants were asked to connect the numbers in order as quickly as possible. A maximum time of 300 seconds was allowed before discontinuing the test. Direct scores of TMT-A were the time in seconds taken to complete task.
executive function assessed by TMT-A | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  The trail marking test A (TMT-A): The TMT-A consisted of a standardized page on which the numbers 1 to 25 are scattered within circles, and the participants were asked to connect the numbers in order as quickly as possible. A maximum time of 300 seconds was allowed before discontinuing the test. Direct scores of TMT-A were the time in seconds taken to complete task.
executive function assessed by DSST | Before the intervention
  Digit Symbol Substitution Test (DSST): The DSST was used to assess visual search, and perceptual and graphomotor speed. The number of correct substitutions during a 90-second interval was used as the score.
executive function assessed by DSST | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  Digit Symbol Substitution Test (DSST): The DSST was used to assess visual search, and perceptual and graphomotor speed. The number of correct substitutions during a 90-second interval was used as the score.
concentration function assessed by DST | Before the intervention
  Digit Span Test (DST): including digit span forwards (DSF) and digit span backwards (DSB)
concentration function assessed by DST | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  Digit Span Test (DST): including digit span forwards (DSF) and digit span backwards (DSB)
quality of life assessed by the Barthel index | Before the intervention
  Barthel index:The main aim is to establish degree of independence from any help, physical or verbal, however minor and for whatever reason.
quality of life assessed by the Barthel index | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  Barthel index:The main aim is to establish degree of independence from any help, physical or verbal, however minor and for whatever reason.
quality of life assessed by EQ-5D-5L | Before the intervention
  European quality of life-5 dimensions with 5 level (EQ-5D-5L): The descriptive system of the EQ-5D comprises five dimensions: mobility (MO), self-care (SC), usual activities (UA), pain/discomfort (PD), and anxiety/depression (AD); each dimension is described at five levels, corresponding roughly to no, slight, moderate, severe, and extreme problems.
quality of life assessed by EQ-5D-5L | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  European quality of life-5 dimensions with 5 level (EQ-5D-5L): The descriptive system of the EQ-5D comprises five dimensions: mobility (MO), self-care (SC), usual activities (UA), pain/discomfort (PD), and anxiety/depression (AD); each dimension is described at five levels, corresponding roughly to no, slight, moderate, severe, and extreme problems.
quality of life assessed by IADL | Before the intervention
  The Lawton instrumental activities of daily living scale (IADL): IADL is an appropriate instrument to assess independent living skills. The instrument is most useful for identifying how a person is functioning at the present time, and to identify improvement or deterioration over time. There are eight domains of function measured with the Lawton IADL scale. Women are scored on all 8 areas of function; historically, for men, the areas of food preparation, housekeeping, laundering are excluded. Clients are scored according to their highest level of functioning in that category. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men.
quality of life assessed by IADL | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  The Lawton instrumental activities of daily living scale (IADL): IADL is an appropriate instrument to assess independent living skills. The instrument is most useful for identifying how a person is functioning at the present time, and to identify improvement or deterioration over time. There are eight domains of function measured with the Lawton IADL scale. Women are scored on all 8 areas of function; historically, for men, the areas of food preparation, housekeeping, laundering are excluded. Clients are scored according to their highest level of functioning in that category. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men.
quality of life assessed by PSMS | Before the intervention
  Physical Self-Maintenance Scale (PSMS): To assess functional abilities in elderly patients. The format the PSMS is first a six item based on the ADL and then eight-items based on the IADL scale. A 5-point scale for responses ranges from total independence to total dependence.
quality of life assessed by PSMS | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  Physical Self-Maintenance Scale (PSMS): To assess functional abilities in elderly patients. The format the PSMS is first a six item based on the ADL and then eight-items based on the IADL scale. A 5-point scale for responses ranges from total independence to total dependence.
quality of life assessed by SF-36 | Before the intervention
  The short-form 36 item health survey (SF-36): The SF-36 includes one multi-item scale that assesses eight health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions.
quality of life assessed by SF-36 | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  The short-form 36 item health survey (SF-36): The SF-36 includes one multi-item scale that assesses eight health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions.
social support assessed by SSRS | Before the intervention
  Social Support Rating Scale (SSRS): SSRS developed by Xiao was utilized to measure social support. The 10-item scale consists of 3 dimensions including objective support, subjective support and availability. Higher scores indicate higher levels of social support. The scale has presented impressive validity and reliability in Chinese population.
social support assessed by SSRS | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  Social Support Rating Scale (SSRS): SSRS developed by Xiao was utilized to measure social support. The 10-item scale consists of 3 dimensions including objective support, subjective support and availability. Higher scores indicate higher levels of social support. The scale has presented impressive validity and reliability in Chinese population.
quality of sleep assessed by PSQI | Before the intervention
  Pittsburgh sleep quality index (PSQI): Sleep quality was assessed using the Chinese version of the PSQI, which is composed of 19 items classified into seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction during the past month. Each component is weighted from 0 to 3, generating one global score ranging from 0 to 21. The higher score the poorer sleep quality.
quality of sleep assessed by PSQI | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  Pittsburgh sleep quality index (PSQI): Sleep quality was assessed using the Chinese version of the PSQI, which is composed of 19 items classified into seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction during the past month. Each component is weighted from 0 to 3, generating one global score ranging from 0 to 21. The higher score the poorer sleep quality.
emotion assessed by GDS-15 | Before the intervention
  Geriatric Depression Scale (GDS-15): The short form including 15 items. Items represent characteristics of depression in the elderly in the affective (e.g., sadness, apathy, crying) and cognitive domains (e.g., thoughts of hopelessness, helplessness, guilt, worthlessness. Higher GDS scores are indicative of more severe depression.
emotion assessed by GDS-15 | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  Geriatric Depression Scale (GDS-15): The short form including 15 items. Items represent characteristics of depression in the elderly in the affective (e.g., sadness, apathy, crying) and cognitive domains (e.g., thoughts of hopelessness, helplessness, guilt, worthlessness. Higher GDS scores are indicative of more severe depression.
cognitive function assessed by The Montreal Cognitive Assessment (MoCA) | Before the intervention
  The MoCA is a 1-page test that measures several cognitive domains (visual perception, executive skills, language, attention, memory and orientation). The MoCA score ranges from 0 to 30 (30 = best) and was chosen for its relatively high sensitivity for mild cognitive impairment.
cognitive function assessed by The Montreal Cognitive Assessment (MoCA) | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  The MoCA is a 1-page test that measures several cognitive domains (visual perception, executive skills, language, attention, memory and orientation). The MoCA score ranges from 0 to 30 (30 = best) and was chosen for its relatively high sensitivity for mild cognitive impairment.

OTHER OUTCOMES:
MRI--T1-weighted structure imaging | Before the intervention
  For the T1 MRI images, we first performed quality control using CAT12 to exclude subjects with quality scores lower than "B". Next, we used the recon-all command of FreeSurfer 6.0.0 for brain extraction, tissue segmentation, cortical reconstruction, and brain region labeling for each subject's brain images. We extracted the thickness, surface area, volume for cortical structures, and volume of subcortical structures in different brain regions based on the DK+Aseg parcellation template. Finally, the brain images of each subject were nonlinearly aligned to the MNI152 template using ANTs alignment toolkit for subsequent analysis of BOLD fMRI and DWI images.
MRI--T1-weighted structure imaging | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  For the T1 MRI images, we first performed quality control using CAT12 to exclude subjects with quality scores lower than "B". Next, we used the recon-all command of FreeSurfer 6.0.0 for brain extraction, tissue segmentation, cortical reconstruction, and brain region labeling for each subject's brain images. We extracted the thickness, surface area, volume for cortical structures, and volume of subcortical structures in different brain regions based on the DK+Aseg parcellation template. Finally, the brain images of each subject were nonlinearly aligned to the MNI152 template using ANTs alignment toolkit for subsequent analysis of BOLD fMRI and DWI images.
MRI--resting functional MRI (rfMRI) imaging | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  We used the alignment results of the T1-weighted image of each subject to transform the resting-state images into MNI152 space , and calculated the functional connectivity between all brain regions, as well as the ALFF, fALFF mean values for each brain region according to the DK+Aseg partitioning template.
MRI--resting functional MRI (rfMRI) imaging | Before the intervention
  We used the alignment results of the T1-weighted image of each subject to transform the resting-state images into MNI152 space , and calculated the functional connectivity between all brain regions, as well as the ALFF, fALFF mean values for each brain region according to the DK+Aseg partitioning template.
MRI--diffusion-weighted imaging (DWI). | Before the intervention
  For DWI images, we mainly used the FSL toolkit for processing. First, the b0 images of each subject were aligned with the T1 images, followed by eddy correction and head motion correction, and detection and replacement of outliers. Next, we used the DK+Aseg parcellation template for probabilistic fiber tracking of DWI images for each subject, and finally generated a probabilistic white matter connectivity matrix for each brain region for subsequent extraction of graph theoretical metrics.
MRI--diffusion-weighted imaging (DWI). | 6 weeks, 12 weeks,3 months, 6 months, 12 months after the intervention
  For DWI images, we mainly used the FSL toolkit for processing. First, the b0 images of each subject were aligned with the T1 images, followed by eddy correction and head motion correction, and detection and replacement of outliers. Next, we used the DK+Aseg parcellation template for probabilistic fiber tracking of DWI images for each subject, and finally generated a probabilistic white matter connectivity matrix for each brain region for subsequent extraction of graph theoretical metrics.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wang, professor, Study Chair — Deputy Director, Professor, School of Public Health, Fudan University
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No